CLINICAL TRIAL: NCT02592213
Title: Treatment of Breast Cancer Related Lymphedema With Cell-assisted Lipotransfer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Navid Toyserkani, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-20150109
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment of lymphedema with cell-assisted lipotransfer using autologous stromal vascular fraction
  Interventions: Procedure: Cell-assisted lipotransfer

INTERVENTIONS:
Procedure: Cell-assisted lipotransfer — Stromal vascular fraction, autologous. Isolated using Celution System (Cytori)

SUMMARY:
Breast cancer is the most common cancer type among women. Treatment in many cases involves axillary lymphadenectomy followed by radiation therapy. This increases the risk of lymphedema development which occurs in up to 30% of such cases. The present treatment paradigm is conservative with compression garments. There is a need for more effective treatment options and regenerative medicine offers hope for a change to a more curative approach. This Phase 2 trial will examine the efficacy and safety of treatment with freshly isolated adipose-derived stromal cells administered as a cell-assisted lipotransfer to the affected axillary region.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer type among women. Treatment in many cases involves axillary lymphadenectomy followed by radiation therapy. This increases the risk of lymphedema development which occurs in up to 30% of such cases. The present treatment paradigm is conservative with compression garments. There is a need for more effective treatment options and regenerative medicine offers hope for a change to a more curative approach. This Phase 2 trial will examine the efficacy and safety of treatment with freshly isolated adipose-deried stromal cells administered as a cell-assisted lipotransfer to the affected axillary region.

Investigators plan to include 10 patients with unilateral lymphedema after previous breast cancer treatment

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral arm lymphedema secondary to breast cancer treatment including lymph node dissection.
2. The patient understands the nature and purpose of this study and the study procedures and has signed informed consent.
3. The opposite upper extremity is healthy.
4. ASA score of 1 or 2.
5. The patient is able to read, understand, and complete Danish questionnaires.
6. Lymphedema grade 1 or 2. A minimum circumference distance of 2cm on either lower or upper arm.

Exclusion Criteria:

1. The patient is pregnant or lactating.
2. The patient has bilateral lymphedema of the upper extremities.
3. The patient has or has had other malignancies other than breast cancer.
4. The patient is treated with anti-diabetic medication.
5. The patient is diagnosed with any form of psychotic disorder.
6. The patient is smoking.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in arm volume | Baseline, 1, 3, 6, 12 and 48 months
  Assessed by clinical measurements

SECONDARY OUTCOMES:
Side effects of treatment | 1, 3, 6, 12 and 48 months
  Any side effects of experimental treatment. Assessed by asking the patient at each visit. All reported findings will be reported at study completion
Subjective change assessed LYMQOL questionnaire | Baseline, 1, 3, 6, 12 and 48 months
  Subjective change of lymphedema assessed by questionnaire
Subjective change assessed DASH questionnaire | Baseline, 1, 3, 6, 12 and 48 months
  Subjective change of lymphedema assessed by questionnaire
Change in lymph drainage | Baseline and 12 months
  Change in lymph drainage assessed by lymphoscintigraphy compared with preoperative lymphoscintigraphy
Subjective change in feeling of tension in arm assessed by numeric scale from 0-10 | Baseline, 1, 3, 6, 12 and 48 months
  Feeling of tension in the arm (separately) 0=healthy and 10=worst imaginable
Subjective change in feeling of heaviness in arm assessed by numeric scale from 0-10 | Baseline, 1, 3, 6, 12 and 48 months
  Feeling of heaviness in the arm (separately) 0=healthy and 10=worst imaginable
Change in arm volume | Baseline, 3, 6 and 12 months
  Assessed by DXA scan
Number of arm infections | Baseline, 1, 3, 6, 12 and 48 months
  Number of arm infections needing antibiotic treatment. Assesed by asking the patient each visit.
Change in conservative lymphedema treatment | Baseline, 1, 3, 6, 12 and 48 months
  Change in use or type of conservative lymphedema treatments. Assesed by asking the patient each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Navid M Toyserkani, MD, Principal Investigator — Dept. Plastic and Reconstructive Surgery, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Toyserkani NM, Jensen CH, Andersen DC, Sheikh SP, Sorensen JA. Treatment of Breast Cancer-Related Lymphedema with Adipose-Derived Regenerative Cells and Fat Grafts: A Feasibility and Safety Study. Stem Cells Transl Med. 2017 Aug;6(8):1666-1672. doi: 10.1002/sctm.17-0037. Epub 2017 Jun 27. PMID 28653440
- [Derived] Toyserkani NM, Jensen CH, Sheikh SP, Sorensen JA. Cell-Assisted Lipotransfer Using Autologous Adipose-Derived Stromal Cells for Alleviation of Breast Cancer-Related Lymphedema. Stem Cells Transl Med. 2016 Jul;5(7):857-9. doi: 10.5966/sctm.2015-0357. Epub 2016 May 5. PMID 27151914